CLINICAL TRIAL: NCT06685510
Title: The Relation Between the Prognosis of Subthalamic Nucleus Deep Brain Stimulation Surgery by Microlesion Effect and Electrode Position
Acronym: Microlesion Ef
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: LC23DBSIIT-HW02
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease (PD); Deep Brain Stimulation
Keywords: Parkinson's disease; Microlesion Effect; Functional Neuroimages; Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: the score of UPDRS item — The score of MDS-UPDRS item 3.1 greater or equal to 2 during the drug-off period at baseline
Other: the score of UPDRS item — The score of MDS-UPDRS item 3.3 greater or equal to 2 during the drug-off period at baseline
Other: the score of UPDRS item — The score of MDS-UPDRS item 3.10 greater or equal to 2 during the drug-off period at baseline
Other: the score of UPDRS item — Any one of the MDS UPDRS 3.15-3.17 scores greater or equal to 2 during the drug-off period at baseline
Other: the score of UPDRS item — Sum of MDS UPDRS 4.1-4.2 scores greater than or equal to 3

SUMMARY:
BACKGROUND: Parkinson's disease (PD) is a common movement disorder whose main symptoms include resting tremor, rigidity and bradykinesia. Deep Brain Stimulation (DBS) has become one of the most effective treatments for PD by implanting electrodes in specific deep brain nuclei to alleviate motor symptoms in PD patients. During the implantation of electrodes in the DBS procedure, small lesions produced are known as the Microlesion Effect, which disappears within a short period. The MLE efficacy is positively correlated with the overall efficacy of DBS, but whether the MLE efficacy is affected by the symptoms has not yet been investigated, and a large-sample study is needed to further validate this. This study aims to examine the relationship between electrode implantation location and the prediction of MLE efficacy produced by STN-DBS surgery in PD patients, assess the correlation between electrode implantation location and DBS efficacy in PD patients, and analyze the role of brain networks in the process. The study will also analyze the relationship between micro-destructive effects and long-term DBS efficacy, providing more effective efficacy prediction and a more accurate selection of electrode implantation locations for DBS treatment in PD patients. This study will guide the clinical practice of DBS treatment in PD patients and provide an important reference for future research in related fields.

Object: Primary Parkinson's Disease patients between the ages of 18 and 75 years who meet STN-DBS surgery criteria Aim: To observe the relationship between predicted efficacy and implantation location of STN-DBS for MLE in PD surgery

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson Disease
2. Age from 18 to 80 years old
3. Performed bilateral STN-DBS

Exclusion Criteria:

1. Does not meet STN-DBS surgical criteria
2. Patients with severely offset electrode implantation position (imaging)
3. Not fulfilling the criteria for an arbitrary cohort under exposure conditions;
4. Patients who are unable to voluntarily sign an informed consent form;
5. Patients who do not agree to cooperate with follow-up visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic Parkinson's disease patients who consecutively consulted the Second Affiliated Hospital of Nanchang University's PD-specialized outpatient clinic were collected as the subjects.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparing MLE and DBS efficacy | From baseline to 24 hours, 48 hours, 7 days ,6 months,one year after surgery
  Based on the improvement rate of short-term postoperative MDS UPDRS-III scores compared with baseline MDS UPDRS-III scores, three subgroups were divided within each cohort into the <20% group, the 20%-40% group, and the >40% group. General statistical analyses of MDS UPDRS-III scores were performed for each subgroup within each cohort, and the mean and standard deviation were calculated. Pearson correlation coefficient analysis was performed on the MDS UPDRS-III score data. Data on MDS UPDRS-III scores of different subgroups within different cohorts were normalized to include short-term postoperative MDS UPDRS-III scores as an independent variable and postoperative post-start-up MDS UPDRS-III scores as a dependent variable, and to include baseline period, postoperative post-start-up, postoperative 6-months, and 12-months MDS UPDRS-III score as a covariate, ANCOVA was performed to observe the differences and correlations of each data node.

SECONDARY OUTCOMES:
Comparison of the efficacy of electrode positions in relation to different positions of the nucleus pulposus | From baseline to 24 hours, 48 hours, 7 days ,6 months,one year after surgery
  Electrode position reconstruction was performed on all subject imaging data. Improvement rates and mean improvement rates were calculated for MDS UPDRS-III scores in the short-term postoperative period, after postoperative start-up, and at 6 and 12 months postoperatively compared to baseline. MLE regional analyses were performed for each subgroup within each cohort, electrode position efficacy heat maps were calculated, and the heat maps were qualitatively analyzed to discuss the relationship between electrode position and efficacy.
Compare short-term postoperative efficacy with postoperative efficacy after start-up | From baseline to 24 hours, 48 hours, 7 days ,6 months,one year after surgery
  Improvement rates within the cohort were calculated and analyzed with general statistics for short-term postoperative, postoperative boot-up, and postoperative 6-month and 12-month comparisons of baseline MDS UPDRS-III scores, and the mean and standard deviation of the improvement rates within the cohort for postoperative boot-up, and postoperative 6-month and 12-month comparisons of baseline PDQ-39 scores were calculated. Differences in improvement rate mean at each time point within the cohort were compared, and linear regression analyses of improvement rates were performed to qualitatively analyze the relationship between short-term postoperative outcomes and long-term postoperative outcomes after postoperative start-up and postoperatively.
Compare the difference in the rate of improvement in MDS UPDRS-III scores within the postoperative pre-opening period | From baseline to 24 hours, 48 hours, 7 days ,6 months,one year after surgery
  General statistical analyses of MDS UPDRS-III scores within the cohort, subgroups within the cohort, and subgroups within the subgroups and improvement rates compared to baseline were performed to compare the differences in data between cohorts, subgroups, and subgroups within the cohort, and Pearson's correlation analysis, analysis of variance (ANOVA), and qualitative analyses were used to look at the efficacy of postoperative MLE.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang L, Zhao J, Wang H, Chen L, Shi Q, Yang X, Ma H, Zhu Y, Li Z, Huang W. The microlesion effect is associated with global cognitive impairment and predicts motor outcomes after subthalamic deep brain stimulation in Parkinson's disease. J Neurol. 2025 Oct 18;272(11):708. doi: 10.1007/s00415-025-13443-z. PMID 41109904